CLINICAL TRIAL: NCT05321719
Title: Multi-Media Parent-based Intervention to Promote Dental Hygiene Among Young Children: BeReady2Smile
Brief Title: Multi-Media Parent-based Intervention to Promote Dental Hygiene Among Young Children: BeReady2Smile II
Acronym: BR2S-II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Research Behavioral Intervention Strategies, Inc. (Industry)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: DE027001-02; 5R44DE027001-03 (NIH)
Record Dates: First submitted 2022-01-26; First posted 2022-04-11 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Plaque
MeSH Terms: conditions — Plaque, Amyloid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental: BeReady2Smile Video, App, & Coach (Experimental): This arm will test the feasibility of the BeReady2Smile Video and App to promote dental health of young children with a parent education program.
  Interventions: Behavioral: Comparison Condition
- Assess the Contributions of BRS2 Components (Experimental): Outcomes of video, app, and coach
  Interventions: Behavioral: BeReady2Smile video only; Behavioral: BeReady2Smile video and BeReady2Smile app completely self-guided; Behavioral: "Complete" BeReady2Smile video and BeReady2Smile app guided by a Coach

INTERVENTIONS:
Behavioral: Comparison Condition — In this Phase II project, BR2S will be evaluated for efficacy relative to a usual care control. Investigators expect BR2S to improve outcomes on behavioral change, self-efficacy, establishment of a dental home, knowledge, and attitudes in real settings relative to the usual care condition. The outcome measures include a direct clinical dental measure as well as observational measures of parental behavior. The study will also provide important information regarding the various types and combinations of BeReady2Smile product components for dissemination. The long-term goal of the program is to help parents provide the foundation for a lifetime free from preventable oral disease.
  Arms: Experimental: BeReady2Smile Video, App, & Coach
Behavioral: BeReady2Smile video only — The video will be viewed at the Head Start site after informed consent and T1 questionnaires and plaque assessment. The video will include concrete demonstrations and feature diversity in settings and actors in video content derived from actual peer-based parenting education sessions. Parents' ability to "see themselves" in the content makes them more likely to engage in discussions about dental health. Supporting these conversations has been identified as an important need. For example, in a recent environmental scan prepared by the Association of State and Territorial Dental Directors the lack of communication strategies was identified as a gap in oral health educational resources. Specifically mentioned was the lack of oral health curricula that support interactive communication between families and home visitors. Families struggle with such dialogues.
  Arms: Assess the Contributions of BRS2 Components
Behavioral: BeReady2Smile video and BeReady2Smile app completely self-guided — In addition to the BeReady2Smile video as described above, the BeReady2Smile app includes: (a) presentation of concepts, behaviors, and examples via video and text, (b) electronically presented check-in questions recorded to a database for review, (c) capture of a 5-minute video of parent-child interactions uploaded for later review by the parent, using a mobile application, (d) daily dental activities (homework), and (e) program feedback recorded to the database. BeReady2Smile will be designed such that before the parent can go on to a new area of learning, the parent must complete the previous lesson. Participants can go back and review previous material in a non-linear format. The database and log-files record all computer activities to track use of each intervention component.
  Arms: Assess the Contributions of BRS2 Components
Behavioral: "Complete" BeReady2Smile video and BeReady2Smile app guided by a Coach — In addition to the BeReady2Smile video and BeReady2Smile app described above, the "complete" intervention includes support via phone and text from a trained facilitator/coach who builds supportive one-on-one relationships with the parent and gives feedback on parent-recorded videos of parent-child interactions of tooth-brushing, designed to facilitate learning and promote engagement with their oral health professional; and tools to create a long-term follow-up plan. Dental behaviors will be tailored for children's developmental level (e.g. twice daily tooth brushing for preschoolers and limiting sugar sweetened beverages or milk in bottles at bed for infants).
  Arms: Assess the Contributions of BRS2 Components

SUMMARY:
"BeReady2Smile (BR2S)", based on successful results from the Phase I SBIR feasibility/usability research of the prototype, is a coordinated oral health prevention intervention program that provides empirically-supported behavioral parent training (BPT) skills and oral health instruction through the use of video and mobile/web- application. In this Phase II project, BR2S will be evaluated for efficacy relative to a usual care control. The investigators expect BR2S to improve outcomes on behavioral change, self-efficacy, establishment of a dental home, knowledge, and attitudes in real settings relative to our usual care condition. The outcome measures include a direct clinical dental measure as well as observational measures of parental behavior.

The study will also provide important information regarding the various types and combinations of BeReady2Smile product components for dissemination. The long-term goal of the program is to help parents provide the foundation for a lifetime free from preventable oral disease.

DETAILED DESCRIPTION:
Primary Objective: Assess the efficacy of the BR2S intervention program in the context of established parenting education systems (e.g., Head Start and Oregon Parenting Education Collaborative). A sub-sample of participants will complete an observational interaction procedure as measured by The Dyadic Parent-Child Interactive Coding System.

Secondary Objectives:

1. Assess relative contribution of BR2S components to outcomes to provide insight on options for dissemination using Usual Care Video only (UC control) or BeReady2Smile Video only or BeReady2Smile video + app or BeReady2Smile Video + app + coach.
2. Assess aspects of user experience with the BR2S program

Primary Endpoint: This study will provide outcomes for a primary endpoints that will compare BeReady2Smile to comparison (usual care video) as measured by the Plaque Control Record. The Plaque Control Record is a very simple percentage or score of the total amount of bacteria present in the mouth. A tooth has 4 surfaces at the gum line being; the cheek side, tongue side, front side, and back side. A hygienist will disclose or stain up the Bacterial Plaque to show where one may be missing.

Secondary Endpoints: 1. With this study's data, additional secondary endpoints the investigators will investigate the effects of BeReady2Smile video alone and BeReady2Smile video + app compared to the usual-care video as well as the impact of a coach (Oral Health Educator). The investigators will also measure behavioral change, self-efficacy, establishment of dental home knowledge, and attitudes. 2. User experience will be measured by Coach Feedback, App feedback, and Video satisfaction.

Study Population: Caregivers, who have a child 0-6 years, enrolled in a participating social service agency providing parenting education, such as Head Start; and are able to communicate in English or Spanish.

Phase* or Stage: 2

Description of Sites/Facilities Enrolling Participants: The study is being conducted at ORBIS, where the investigators, and bachelor- and masters-level recruitment staff, computer programmers, data management staff, and data analyst are housed. Enrollment of eligible parents, technological adaptations for the intervention, data analysis, and manuscript production will be completed there.

Agency staff at Head Start and Oregon Parenting Education Collaborative will inform parents about the project and will get parent permission to share their contact information with the family recruiters at ORBIS.

Description of Study Intervention/Experimental Manipulation: BR2S is a coordinated oral health prevention intervention program to promote dental health targeted at parents of young children attending parenting education classes and families receiving home visiting services through Head Start. Participants will be randomized in one of 4 experimental conditions (Usual care video; BR2S video; BR2S video + app; BR2Svideo + app + coach) with the primary comparison being between those who were exposed to one or more component of BR2S and those who received a usual care video.

ELIGIBILITY:
Inclusion Criteria:

• Have a child 0-6 years enrolled in a participating social service agency providing parent education, such as Head Start; be able to communicate in English or Spanish.

Exclusion Criteria: Individuals who meet the following criteria will be excluded from the study:

* Parental psychosis or other major mental illness or cognitive disability that would interfere with meaningful participation
* Babies without teeth
* Children with allergies to food dye.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 228 (Actual)
Dates: Start 2023-04-10 (Actual); Primary Completion 2024-04-24 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Change in parental attitudes towards child tooth brushing and caries | T1 (Baseline) and T3 (three month)
  Four scales are included in the questionnaire that were developed for the international study of Adair and colleagues. Included in this study were:
  1. 'Importance and Intention to Brush Child's Teeth' (five items),
  2. 'Parental Efficacy in Relation to Child Tooth brushing' (6 items),
  3. 'Perceived Seriousness of Tooth Decay in Children' (seven items) and
  4. 'Chance Control - Decay Occurs by Chance' (5 items). Response options range from 'strongly agree' (=1) to 'strongly disagree' (=5).

SECONDARY OUTCOMES:
Knowledge | T1 (Baseline) and T3 (three month)
  As part of the pre- and post-intervention questionnaires, parents will complete a 15-item knowledge inventory of young children's oral health. The items include recommendations for home hygiene and dental health (nine items), statements about the caries process (two items) and dental development (three items). For each item, parents indicated their level of knowledge as 'didn't know', 'sorta know' and 'know for sure'; item scoring ranges from 1 to 3 points, respectively.
Parents' confidence in brushing | T1 (Baseline) and T3 (three month)
  Investigators will use a Likert scale to determine parents' confidence in brushing their child's teeth twice a day. The question asked was 'If you already don't brush twice a day, how confident are you that, if you decided to, you could brush your child's teeth twice (or almost always twice) a day?' Parents responded on a scale of 1-10 how motivated they are to change this behavior.
Connection to Dental Services "Dental Home" | T1 (Baseline) and T3 (three month)
  The dental home concept has been by the American Academy of Pediatric Dentistry that states, "the dental home is the ongoing relationship between the dentist and the patient, inclusive of all aspects of oral health care delivered in a comprehensive, continuously accessible, coordinated, and family-centered way." This concept is intimately linked to a cluster of additional progressive policies currently being advanced by pediatric dentistry including the age one dental visit, outreach to Head Start populations, updating state Medicaid periodicity schedules, and refining clinical care through risk assessment and risk-based interventions. Parents will be asked to provide past dental services to ascertain the presence of an ongoing relationship with a dentist.
Clinical Dental Exam for Plaque | T1 (Baseline) and T3 (three month)
  Children of parents participating in the research will be administered the Plaque Control Record by a Dental Hygienist. The Plaque Control Record was developed to give the therapist, hygienist, or dental educator a simple method of recording the presence of the plaque on individual tooth surfaces: (a) Mesial, (b) Distal (d) Buccal and (d) Lingual. At the exam, a suitable disclosing solution such as Bismarck Brown, Diaplac or similar is painted on all exposed tooth surfaces. After the patient has rinsed, the hygienist (using an explorer or a tip of a probe) examines each stained surface for soft accumulations at the dentogingival junction and are recorded by making a dash in the appropriate spaces on the record form. Those surfaces, which do not have soft accumulations at the dentogingival junction, are not recorded. The index is calculated by dividing the number of plaque containing surfaces by the total number of available surfaces.
Usage of Application | Once a week through study completion at 12 weeks
  Throughout the clinical trial all participant activity both online and through the app will be recorded to a MySQL database. Process indicants of acceptability included the following indices of participation: (1) attrition; (2) session completion; and (3) extent of intervention participation (e.g., time online).
Satisfaction of Video and App | T2 (one month) and T3 (three month)
  Parents will rate the video and app on a 4-point scale from 1="not at all" (negative) to 4="Very" (positive). Parents were asked questions such as "How reasonable did you find the Video", "How much did you like the video for learning information taught", "How clear was information taught", "How useful did you find BeReady2Smile" and "I would recommend the BR2S video to other parents".
Direct observation of Parenting Behavior | T1 (Baseline) and T3 (three month)
  An observational assessment of parenting behavior during mother-child interactions, consisting of three 5-min tasks, tooth brushing, a child-led play session, and a parent-led play session/clean-up task. The interactions were coded using the Dyadic Parent-Child Interaction Coding System (Eyberg, et al., 2013). Coders were blind to group and assessment period, and 20% of interactions were double coded for reliability purposes.

CONTACTS AND LOCATIONS:
Overall Officials: David R Smith, PhD, Principal Investigator — Oregon Research Behavioral Intervention Strategies, Inc.
Locations (1):
- Oregon Research Behavioral Intervention Strategies, Inc., Springfield, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] American Academy on Pediatric Dentistry Council on Clinical Affairs. Policy on early childhood caries (ECC): unique challenges and treatment option. Pediatr Dent. 2008-2009;30(7 Suppl):44-6. No abstract available. PMID 19216382
- [Background] Section On Oral Health. Maintaining and improving the oral health of young children. Pediatrics. 2014 Dec;134(6):1224-9. doi: 10.1542/peds.2014-2984. PMID 25422016
- [Background] Barkley RA. Attention-deficit/hyperactivity disorder, self-regulation, and time: toward a more comprehensive theory. J Dev Behav Pediatr. 1997 Aug;18(4):271-9. PMID 9276836
- [Background] Brinkmeyer, M., & Eyberg, S. M. (2003). Parent-child interaction therapy for oppositional children. In A.E. Kazdin & J. R. Weisz (Eds.), Evidence-based psychotherapies for children and adolescents (pp. 204-223). New York: Guilford.
- [Background] Forgatch, M. S., & Patterson, G. R. (2010). Parent Management Training -- Oregon Model: An intervention for antisocial behavior in children and adolescents. In J. R. Weisz & A. E. Kazdin (Eds.), Evidence based psychotherapies for children and adolescents (2nd ed., pp. 159-178). New York, NY: Guilford.
- [Background] Huebner CE, Riedy CA. Behavioral determinants of brushing young children's teeth: implications for anticipatory guidance. Pediatr Dent. 2010 Jan-Feb;32(1):48-55. PMID 20298653
- [Background] Kazdin AE. Evidence-based treatment and practice: new opportunities to bridge clinical research and practice, enhance the knowledge base, and improve patient care. Am Psychol. 2008 Apr;63(3):146-59. doi: 10.1037/0003-066X.63.3.146. PMID 18377105
- [Background] Pine CM, Adair PM, Petersen PE, Douglass C, Burnside G, Nicoll AD, Gillett A, Anderson R, Beighton D, Jin-You B, Broukal Z, Brown JP, Chestnutt IG, Declerck D, Devine D, Espelid I, Falcolini G, Ping FX, Freeman R, Gibbons D, Gugushe T, Harris R, Kirkham J, Lo EC, Marsh P, Maupome G, Naidoo S, Ramos-Gomez F, Sutton BK, Williams S. Developing explanatory models of health inequalities in childhood dental caries. Community Dent Health. 2004 Mar;21(1 Suppl):86-95. PMID 15072477
- [Background] Webster-Stratton, C., & Reid, M. J. (2003). Strengthening social and emotional competence in young children--the foundation for early school readiness and success: Incredible Years Classroom Social Skills and Problem-Solving curriculum. Infants and Young Children, 17(2), 96-113.
- [Background] Adair PM, Pine CM, Burnside G, Nicoll AD, Gillett A, Anwar S, Broukal Z, Chestnutt IG, Declerck D, Ping FX, Ferro R, Freeman R, Grant-Mills D, Gugushe T, Hunsrisakhun J, Irigoyen-Camacho M, Lo EC, Moola MH, Naidoo S, Nyandindi U, Poulsen VJ, Ramos-Gomez F, Razanamihaja N, Shahid S, Skeie MS, Skur OP, Splieth C, Soo TC, Whelton H, Young DW. Familial and cultural perceptions and beliefs of oral hygiene and dietary practices among ethnically and socio-economicall diverse groups. Community Dent Health. 2004 Mar;21(1 Suppl):102-11. PMID 15072479
- [Background] Huebner CE, Milgrom P. Evaluation of a parent-designed programme to support tooth brushing of infants and young children. Int J Dent Hyg. 2015 Feb;13(1):65-73. doi: 10.1111/idh.12100. Epub 2014 Jul 29. PMID 25070036
- [Background] Edelstein, B. L. (2008). Environmental factors in implementing the dental home for all young children. National Oral Policy Center at Children's Dental Health Project.
- [Background] American Academy of Pediatric Dentistry reference manual 2007-2008. Pediatr Dent. 2007-2008;29(7 Suppl):1-271. No abstract available. PMID 18268823
- [Background] O'Leary TJ, Drake RB, Naylor JE. The plaque control record. J Periodontol. 1972 Jan;43(1):38. doi: 10.1902/jop.1972.43.1.38. No abstract available. PMID 4500182
- See also: Intervention website — https://beready2smile.com